CLINICAL TRIAL: NCT06836206
Title: The Effect of Gum Arabic (GA) on Adult Dialysis Patients in Abu Dhabi: A Prospective Randomized-controlled Trial (The GADAD Study)
Brief Title: The Effect of Gum Arabic (GA) on Residual Renal Function in Adult Dialysis Patients in Abu Dhabi
Acronym: GAESRD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abu Dhabi Health Services Company (Other Government)
Responsible Party: Principal Investigator, Stephen Geoffrey Holt, SEHA Kidney Care (SKC) Professor Director, Abu Dhabi Health Services Company
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HREC SEHA-IRB- 814
Record Dates: First submitted 2025-01-30; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: End Stage Renal Disease (ESRD)
Keywords: Gum Arabic; ESRD; Acacia seyal and Acacia senegal
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Gum Arabic; Water

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, crossover trial
  Intervention:
  Treatment A: Gum Arabic (Acacia seyal and Acacia senegal) in 100ml water Treatment B: Water 100ml Patients will receive either treatment A or B for 3 months followed by a washout then the other arm of therapy. ie randomized to the treatment sequence AB or BA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A: 30g powdered GA in 100ml water, consumed daily (Experimental): Treatment A: 30g powdered GA in 100ml water, consumed daily
  Interventions: Dietary Supplement: Gum Arabic
- Treatment B: 100ml water, consumed daily. (Other): Treatment B: 100ml water, consumed daily. Participants will follow their usual medications and lifestyle, randomized into two sequences (AB or BA).
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Gum Arabic — Gum Arabic (Acacia seyal and Acacia senegal) 30g powdered GA in 100ml water, consumed daily.
  Arms: Treatment A: 30g powdered GA in 100ml water, consumed daily
Other: Water — 100ml water, consumed daily
  Arms: Treatment B: 100ml water, consumed daily.

SUMMARY:
Gum Arabic (GA), derived from Acacia trees, has shown potential benefits in metabolic, renal, and inflammatory conditions. This study explores the impact of GA on residual renal function in end-stage renal disease (ESRD) patients undergoing dialysis, as current evidence is limited.

DETAILED DESCRIPTION:
Gum Arabic (GA) is an exudate with a gummy texture obtained from Acacia seyal and Acacia senegal. It is an arabinogalactan-protein complex and is composed of magnesium, calcium, and potassium salts of Arabic acid. GA is widely used in sub-Saharan African countries as a traditional remedy for many years. Ingestion of GA has been claimed to have beneficial effects in several health conditions like metabolic syndrome, renal failure, hypertension, gingivitis, anaemia, and hypercholesterolemia. Clinical trials conducted earlier have studied the effect of GA on metabolic disorders like type 2 diabetes mellitus, hyperlipidaemia, gastrointestinal health, oral health, renal diseases, and diseases like sickle cell anaemia and rheumatoid arthritis. A few studies have described GA to exhibit antioxidant properties, anti-inflammatory, probiotic, and antibacterial properties. GA has high fibre content causing satiety and is suggested as a good dietary fibre in patients with chronic kidney disease (CKD) based on its effect on various physiological and biochemical parameters.

The effect of GA on CKD patients has only been studied in a few publications. A study of patients undergoing regular haemodialysis showed supplementation of GA 50g/day along with low protein diet for 3 months resulted in a significant reduction in serum urea, creatinine, uric acid and phosphate levels and a significant increase in serum calcium levels. Another clinical trial conducted in Saudi Arabia among CKD patients showed that supplementing the diet with GA for four weeks significantly reduced C-reactive protein (CRP) levels however, four weeks supplementation did not show any effect on the serum urea and creatinine levels. Another study on forty ESRD patients on haemodialysis showed that GA supplementation of 30g/day for 12 weeks significantly improved Hb levels and augmented total antioxidant capacity whilst reducing CRP. A clinical trial conducted on patients with stage 2 or 3 CKD demonstrated that GA supplementation of 25g/day for a year was well tolerated and was associated with a slowing in the rate of decline of renal function as measured by eGFR. A single case study published in 2009 reported the postponement of dialysis for six years in a young girl with advanced CKD using GA 1-1.5 g/kg/day combined with traditional conservative (dietary and pharmacological) treatments . A systematic review on efficacy and safety of GA in patients with CKD suggested that GA supplementation may improve parameters like serum creatinine, urea, sodium, and potassium, but early-stage intervention and long duration of therapy were more likely to improve renal parameters.

GA is commonly used in the making of food products like puddings, frostings and candies . It has demulcent property for which it is used in medications and is generally recognized as safe by the US Food and Drug Administration. Earlier animal studies in toxicology have shown that there were no significant harmful effects observed on chronic intake of GA and no known teratogenic effects in animals .

There is a paucity of data on drug interactions, but studies have shown that concurrent use of oral GA and amoxicillin changed the pharmacokinetics resulting in a significant reduction in the absorption of amoxicillin leading to sub therapeutic plasma concentrations. A animal study on gastric ulcers demonstrated that GA administration potentiated the anti-ulcer effect of ranitidine.

Limited evidence supports the beneficial effects of oral GA on renal function, and there are no definitive studies demonstrating an improvement in residual renal function in ESRD patients undergoing haemodialysis.

This trial aims to assess the effect of GA on residual renal function in ESRD patients on dialysis.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this trial, an individual must meet all the following criteria:

1. Men and women ≥18 years of age with diagnosed ESRD and prescribed regular dialysis at least once a week, weekly at least for past two weeks.
2. For past two weeks including women of childbearing potential who are currently adopting any method of contraception or have completed the family and undergone sterilization procedures and women of non-childbearing potential.
3. Patients with residual renal function - Patients who produce a minimum of 200 ml of urine during a full day of collection (A full day collection: the patient discards the first urine sample on the day of collection then collects all urine for the entire day and night and collects the first urine sample of the next day) r on a non-dialysis long break day.
4. Able and willing to complete the whole period of the study (maximum of 266 days from enrolment).
5. With the ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the protocol.

Exclusion Criteria:

1. Women of childbearing potential not adopting any methods of contraception, have not undergone sterilization.
2. Women Pregnant or lactating
3. Patients who plan to conceive (or for their partners to conceive) within 12 months of randomization.
4. Patient presenting with serum K+levels ≥ 6mmol/L based on the last two reports as per medical records.
5. Patients who produce less than 200 ml of urine during 24 hours urine collection at baseline assessment.
6. Peritoneal dialysis.
7. Kidney transplant or booked for a live transplant within 259 days of randomization.
8. Patients gaining >4 kg between dialysis sessions in the past 2 weeks.
9. People with known allergies to quillaja bark or similar tree bark.
10. Patients are already participating in another clinical trial (excluding COVID-19 vaccine or COVID-19 drug trials).
11. Patients on immunosuppression for kidney transplant.

Additional exclusion criteria for follow-up visits.

1. Patient informs of pregnancy.
2. Severe adverse reaction to the interventional product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean average clearance of urea and creatinine in a full 24-hour urine collection. | 3 months
  To evaluate the effect of Gum Arabic (GA) on residual renal function in end stage renal disease (ESRD) patients on dialysis as measured by the achievement of at least 5 millilitres/minute improvement in mean average urea creatinine clearance.

SECONDARY OUTCOMES:
Changes in urine volume | 3 months
  Evaluate changes in urine volume collected for 24 hours over long intradialytic period (ml)
Changes in serum lipids | 3 months
  Evaluate changes in serum cholesterol (mmol/l)
Changes in intradialytic weight gain. | 3 months
  Evaluate changes in intradialytic weight gain (kg)
Side effects bad enough to discontinue IP | 3 months
  Percentage of patients who have side effects that cause them to discontinue therapy.(%)
Changes in serum potassium | 3 months
  Serum potassium (mmol/l)

OTHER OUTCOMES:
Exploratory end point | 3 months
  Analyze impacts on cardiac health ECG changes
Exploratory end point | 3 months
  Analyze impacts Fructosamines (mmol/l)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen G Holt, MD, Principal Investigator — Abu Dhabi Health Services Co. -SEHA
Locations (1):
- SEHA Kidney Care (SKC), Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eltayeb IB, Awad AI, Elderbi MA, Shadad SA. Effect of gum arabic on the absorption of a single oral dose of amoxicillin in healthy Sudanese volunteers. J Antimicrob Chemother. 2004 Aug;54(2):577-8. doi: 10.1093/jac/dkh372. Epub 2004 Jul 21. No abstract available. PMID 15269196
- [Background] Collins TF, Welsh JJ, Black TN, Graham SL, O'Donnell MW Jr. Study of the teratogenic potential of guar gum. Food Chem Toxicol. 1987 Nov;25(11):807-14. doi: 10.1016/0278-6915(87)90258-4. PMID 3692386
- [Background] Melnick RL, Huff J, Haseman JK, Dieter MP, Grieshaber CK, Wyand DS, Russfield AB, Murthy AS, Fleischman RW, Lilja HS. Chronic effects of agar, guar gum, gum arabic, locust-bean gum, or tara gum in F344 rats and B6C3F1 mice. Food Chem Toxicol. 1983 Jun;21(3):305-11. doi: 10.1016/0278-6915(83)90065-0. PMID 6683227
- [Background] Al Mosawi AJ. Six-year dialysis freedom in end-stage renal disease. Clin Exp Nephrol. 2009 Oct;13(5):494-500. doi: 10.1007/s10157-009-0181-7. Epub 2009 May 30. PMID 19479191
- [Background] Ali NE, Kaddam LA, Alkarib SY, Kaballo BG, Khalid SA, Higawee A, AbdElhabib A, AlaaAldeen A, Phillips AO, Saeed AM. Gum Arabic (Acacia Senegal) Augmented Total Antioxidant Capacity and Reduced C-Reactive Protein among Haemodialysis Patients in Phase II Trial. Int J Nephrol. 2020 Apr 9;2020:7214673. doi: 10.1155/2020/7214673. eCollection 2020. PMID 32328307
- [Background] Elamin S, Alkhawaja MJ, Bukhamsin AY, Idris MAS, Abdelrahman MM, Abutaleb NK, Housawi AA. Gum Arabic Reduces C-Reactive Protein in Chronic Kidney Disease Patients without Affecting Urea or Indoxyl Sulfate Levels. Int J Nephrol. 2017;2017:9501470. doi: 10.1155/2017/9501470. Epub 2017 May 14. PMID 28589039
- [Background] Ali AA, Ali KE, Fadlalla AE, Khalid KE. The effects of gum arabic oral treatment on the metabolic profile of chronic renal failure patients under regular haemodialysis in Central Sudan. Nat Prod Res. 2008 Jan 10;22(1):12-21. doi: 10.1080/14786410500463544. PMID 17999333
- [Background] Nasir O. Renal and extrarenal effects of gum arabic ( Acacia senegal )--what can be learned from animal experiments? Kidney Blood Press Res. 2013;37(4-5):269-79. doi: 10.1159/000350152. Epub 2013 Aug 11. PMID 24022265
- [Background] Babiker R, Merghani TH, Elmusharaf K, Badi RM, Lang F, Saeed AM. Effects of Gum Arabic ingestion on body mass index and body fat percentage in healthy adult females: two-arm randomized, placebo controlled, double-blind trial. Nutr J. 2012 Dec 15;11:111. doi: 10.1186/1475-2891-11-111. PMID 23241359
- [Background] Jarrar AH, Stojanovska L, Apostolopoulos V, Feehan J, Bataineh MF, Ismail LC, Al Dhaheri AS. The Effect of Gum Arabic (Acacia Senegal) on Cardiovascular Risk Factors and Gastrointestinal Symptoms in Adults at Risk of Metabolic Syndrome: A Randomized Clinical Trial. Nutrients. 2021 Jan 9;13(1):194. doi: 10.3390/nu13010194. PMID 33435475
- [Background] Gafar AM, Ramadan AM, ElSaid NA, Nurelhuda NM. Effect of Gum Arabic on plaque-induced gingivitis: A randomised controlled trial. Saudi Dent J. 2022 Sep;34(6):494-502. doi: 10.1016/j.sdentj.2022.06.002. Epub 2022 Jun 13. PMID 36092515
- [Background] Al-Jubori Y, Ahmed NTB, Albusaidi R, Madden J, Das S, Sirasanagandla SR. The Efficacy of Gum Arabic in Managing Diseases: A Systematic Review of Evidence-Based Clinical Trials. Biomolecules. 2023 Jan 9;13(1):138. doi: 10.3390/biom13010138. PMID 36671523
- [Background] Ashour MA, Fatima W, Imran M, Ghoneim MM, Alshehri S, Shakeel F. A Review on the Main Phytoconstituents, Traditional Uses, Inventions, and Patent Literature of Gum Arabic Emphasizing Acacia seyal. Molecules. 2022 Feb 9;27(4):1171. doi: 10.3390/molecules27041171. PMID 35208961
- [Background] Mayne TJ, Nordyke RJ, Schold JD, Weir MR, Mohan S. Defining a minimal clinically meaningful difference in 12-month estimated glomerular filtration rate for clinical trials in deceased donor kidney transplantation. Clin Transplant. 2021 Jul;35(7):e14326. doi: 10.1111/ctr.14326. Epub 2021 May 5. PMID 33896052
- See also: Gum Arabic in renal disease (GARDS Study): Clinical evidence of dietary supplementation impact on progression of renal dysfunction — https://doi.org/10.1016/j.jff.2021.104515
- See also: Efficacy and Safety of Gum Arabic on Renal Failure Patients: Systematic Review and Meta-analysis — https://www.academia.edu/100913830/Efficacy_and_Safety_of_Gum_Arabic_on_Renal_Failure_Patients_Systematic_Review_and_Meta_analysis
- See also: Al-Yahya AA, Asad M. Antiulcer activity of gum Arabic and its interaction with antiulcer effect of ranitidine in rats. Biomedical Research (India). 2016;27(4). — https://www.alliedacademies.org/articles/antiulcer-activity-of-gum-arabic-and-its-interaction-with-antiulcer-effect-of-ranitidine-in-rats.pdf#